CLINICAL TRIAL: NCT03626168
Title: Bioactive Compounds in Watermelon Modulating Oxidative Stress and Inflammation in Elders: The MOXIE Study
Brief Title: Bioactive Compounds in Watermelon Modulating Oxidative Stress and Inflammation in Elders
Acronym: MOXIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama, Tuscaloosa (Other)
Responsible Party: Principal Investigator, Amy Ellis, Assistant Professor, University of Alabama, Tuscaloosa
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 16MCPRP27260233
Record Dates: First submitted 2018-07-24; First posted 2018-08-10 (Actual); Results first posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Arterial Stiffness; Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: In a double-blind crossover design, women ages 55-69 years were randomized to two 12-ounce servings of 100% watermelon juice per day or an isocaloric placebo for four weeks each with a 2-week washout period in between.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: In this crossover design, the participants principal investigators, and outcomes assessors were blinded as to which treatment (100% watermelon juice or placebo) was consumed at each time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Consumption of 100% watermelon juice (Active Comparator): Consumption of two 12-ounce doses of pasteurized 100% watermelon juice for a four-week period
  Interventions: Dietary Supplement: 100% watermelon juice
- Consumption of a placebo beverage (Placebo Comparator): Consumption of a placebo beverage with comparable sugar content, pH, taste, texture, and color for a four-week period
  Interventions: Other: Placebo beverage

INTERVENTIONS:
Dietary Supplement: 100% watermelon juice — Participants drank two 12-ounce servings of 100% watermelon juice per day for a four-week period.
  Arms: Consumption of 100% watermelon juice
Other: Placebo beverage — Participants drank two 12-ounce servings of a placebo beverage per day for a four-week period.
  Arms: Consumption of a placebo beverage

SUMMARY:
Watermelon is the only food with a unique combination of amino acids and antioxidants that may reduce artery stiffness. However, only 27% of older adults meet the daily recommendation for fruit intake. Because it tastes good and is convenient and easy to consume, watermelon juice is an innovative and impactful intervention to help elders easily meet recommendations for fruit servings. If effective, this intervention would be a simple, inexpensive way to combat cardiovascular diseases (CVD). Results will advance science by providing a better understanding whether four-week consumption of 100% watermelon juice may impact measures of vascular health and inflammation in postmenopausal women.

DETAILED DESCRIPTION:
Purpose and Objectives:

Vascular endothelial dysfunction is an early independent predictor of cardiovascular diseases (CVD), the leading cause of death for women ages 60 and older in the United States1. It is well-known that age-related decreases in vascular endothelial function are partially due to increases in oxidative stress and inflammation.In attempts to combat CVD, previous intervention studies have investigated provision of isolated bioactive food compounds (BFC) in supplemental form. For example, purified lycopene has been shown to decrease oxidative stress, and our previous work supports the supplemental use of glutamine and arginine in improving vascular endothelial function of older adults. Arginine is a precursor for the vasodilatory molecule nitric oxide (NO), and both glutamine and arginine have been shown to attenuate inflammation. Thus, if supplemented together, these compounds would be expected to exert synergist mechanistic effects that improve vascular function.

Watermelon is one of the richest sources of lycopene, and it is among the greatest plant sources of arginine and glutamine. Watermelon also provides high amounts of citrulline (a precursor of arginine) along with the antioxidant ascorbic acid, which enhances the antioxidant and anti-inflammatory effects of carotenoids such as lycopene in biological samples. To date, clinical studies evaluating the potential synergy of these compounds provided by the whole food are lacking on mechanistic and clinical outcomes of CVD. The effects of watermelon supplementation on robust measures of vascular function, inflammation, and oxidative stress in women ages 60 and older are unknown. This study will evaluate the possible impact of multiple bioactive compounds in the natural food matrix of watermelon in order to fully characterize their potential synergy and their influence on CVD risk. Specifically, our proposed study seeks to evaluate the influence of bioactive compounds in 100% watermelon juice, a convenient serving alternative to fresh fruit, using a randomized, double-blind placebo-controlled trial with a crossover design.

Specific Aims:

1. Mechanistic: To determine whether community-dwelling, non-obese women ages 55-69 consuming two 12-ounce servings of 100% watermelon juice per day versus placebo for four weeks will demonstrate:

   1. increases in circulating levels of serum lycopene, citrulline, and arginine using ultra high performance liquid chromatography with photodiode array detector (UPLC-PDA).
   2. improvement in antioxidant status as assessed by the oxygen radical absorbance capacity assay (ORAC) of whole and deproteinated serum
   3. decreases in circulating biomarkers of inflammation Hypotheses: Four-week dietary supplementation with 100% watermelon juice will result in increased antioxidant capacity and decreased inflammation, related to increased serum lycopene, citrulline, and arginine
2. Clinical: To determine whether community-dwelling, women ages 55-69 consuming two 12-ounce servings of 100% watermelon juice per day versus placebo for four weeks will exhibit:

   1. improved vascular endothelial function as assessed by flow-mediated dilation (FMD) and decreased arterial stiffness as assessed by pulse wave analysis (PWA)
   2. decreased low density lipoprotein (LDL) oxidation as assessed by enzyme immunoassay Hypotheses: Four-week dietary supplementation with 100% watermelon juice will result in improved vascular endothelial function, decreased arterial stiffness, and decreased LDL oxidation.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory
* Female
* Age 55-69 years
* Body mass index 18.5 - 29.9 kg/m2 (non-obese)

Exclusion Criteria:

* Food allergy to watermelon
* History of hypotension, chronic hypertension, chronic kidney disease, diabetes, previous cardiac events or procedures, phenylketonuria
* Smoking or other tobacco use
* Use of anticoagulant medications, cholesterol-lowering medications, blood-pressure medications, vasodilatory dietary supplements (garlic, fish oil), or dietary supplements containing lycopene, ascorbic acid, L-glutamine, L-arginine, or L-citrulline
* Weight change > 10% in the previous year

Ages: 55 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2018-05-12 (Actual); Study Completion 2018-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy C Ellis, PhD, RD, Principal Investigator — University of Alabama at Birmingham; Kristi Crowe-White, PhD, RD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ellis AC, Dudenbostel T, Locher JL, Crowe-White K. Modulating Oxidative Stress and Inflammation in Elders: The MOXIE Study. J Nutr Gerontol Geriatr. 2016 Oct-Dec;35(4):219-242. doi: 10.1080/21551197.2016.1250693. PMID 27897608
- [Derived] Ellis AC, Mehta T, Nagabooshanam VA, Dudenbostel T, Locher JL, Crowe-White KM. Daily 100% watermelon juice consumption and vascular function among postmenopausal women: A randomized controlled trial. Nutr Metab Cardiovasc Dis. 2021 Sep 22;31(10):2959-2968. doi: 10.1016/j.numecd.2021.06.022. Epub 2021 Jul 7. PMID 34344546
- [Derived] Crowe-White KM, Voruganti VS, Talevi V, Dudenbostel T, Nagabooshanam VA, Locher JL, Ellis AC. Variation of Serum Lycopene in Response to 100% Watermelon Juice: An Exploratory Analysis of Genetic Variants in a Randomized Controlled Crossover Study. Curr Dev Nutr. 2020 Jun 17;4(7):nzaa102. doi: 10.1093/cdn/nzaa102. eCollection 2020 Jul. PMID 32695957

RESULTS

PARTICIPANT FLOW:
Groups:
- 100% Watermelon Juice First, Then Placebo Beverage: Consumption of two 12-ounce doses of pasteurized 100% watermelon juice for a four-week period
  2-week washout period
  Consumption of two 12-ounce doses of placebo beverage for a four-week period
- Placebo Beverage First, Then 100% Watermelon Juice: Consumption of two 12-ounce doses of placebo beverage for a four-week period
  2-week washout period
  Consumption of two 12-ounce doses of pasteurized 100% watermelon juice for a four-week period
Period: First Intervention (4 Weeks)
Arm/Group | 100% Watermelon Juice First, Then Placebo Beverage | Placebo Beverage First, Then 100% Watermelon Juice
Started | 9 | 12
Completed | 8 | 11
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Began a medication that precluded participation | 0 | 1
Period: Washout (2 Weeks)
Arm/Group | 100% Watermelon Juice First, Then Placebo Beverage | Placebo Beverage First, Then 100% Watermelon Juice
Started | 8 | 11
Completed | 8 | 11
Not Completed | 0 | 0
Period: Second Intervention (4 Weeks)
Arm/Group | 100% Watermelon Juice First, Then Placebo Beverage | Placebo Beverage First, Then 100% Watermelon Juice
Started | 8 | 11
Completed | 8 | 9
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: One participant was randomized, but she began taking a hypertension medication that precluded her participation prior to baseline testing. Three other participants withdrew from the study before completion, but they completed baseline testing.
Groups:
- Placebo Beverage First, Then 100% Watermelon Juice: Consumption of two 12-ounce doses of placebo beverage for a four-week period
  2-week washout period
  Consumption of two 12-ounce doses of 100% watermelon juice for a four-week period
- Total: Total of all reporting groups
Arm/Group | 100% Watermelon Juice First, Then Placebo Beverage | Placebo Beverage First, Then 100% Watermelon Juice | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.78 (4.99) | 58.91 (2.91) | 60.20 (4.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 11 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 11 | 20
Weight [Mean (Standard Deviation); unit: kg] | 59.69 (10.07) | 69.96 (5.75) | 65.34 (9.36)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 22.61 (3.21) | 27.12 (2.51) | 25.08 (3.60)
Serum lycopene [Mean (Standard Deviation); unit: uM] | 1.55 (0.70) | 1.26 (0.87) | 1.37 (0.80)
Serum arginine [Mean (Standard Deviation); unit: uM] | 65.51 (24.54) | 54.64 (16.10) | 58.87 (19.87)
Serum citrulline [Mean (Standard Deviation); unit: uM] | 30.43 (6.82) | 24.23 (6.16) | 26.64 (6.96)
Oxygen radical absorbance capacity (ORAC) [Mean (Standard Deviation); unit: uM Trolox Equivalents] | 642.05 (196.40) | 827.67 (231.07) | 749.51 (231.36)
TNF-alpha [Mean (Standard Deviation); unit: pg/ml] | 2.32 (0.37) | 2.52 (0.56) | 2.44 (0.50)
Oxidized LDL [Mean (Standard Deviation); unit: uM/dl] | 75.10 (12.10) | 75.61 (9.93) | 75.41 (10.48)
Flow-mediated dilation (FMD) [Mean (Standard Deviation); unit: percentage of change in diameter] | 10.17 (7.44) | 7.93 (6.04) | 8.94 (6.62)
Pulse wave velocity (PWV) [Mean (Standard Deviation); unit: meters per second] | 8.40 (0.75) | 8.20 (0.69) | 8.29 (0.71)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Serum Levels of Lycopene at 4 Weeks
Description: Lycopene determined by ultra high performance liquid chromatography with photodiode array detector (UPLC-PDA).
Time Frame: Baseline and 4 Weeks
Population: Serum lycopene was unavailable for one participant due to an insufficient blood sample. With the crossover design, participants completed both arms of the study with a two-week washout period in between.
Measure: Mean (Standard Deviation); unit: uM
Arm/Group | Consumption of 100% Watermelon Juice | Consumption of a Placebo Beverage
Number analyzed (Participants) | 16 | 16
uM | 7.30 (7.55) | 3.09 (4.92)

2. Primary Outcome: Change in Vascular Endothelial Function at 4 Weeks
Description: Determined by brachial artery flow-mediated dilation (FMD). FMD uses ultrasound technology to quantify changes in brachial artery diameter in response to hyperemia. A blood pressure cuff was placed distal to the brachial artery of the right arm with the participant supine and rested. Pre-inflation diameter was recorded for one minute, and the cuff was inflated to 50 mmHg above resting SBP for five minutes. Then, images were recorded for 120 seconds after cuff deflation. Peak diameter was determined as an average of the five highest measurements over five seconds post-deflation. FMD was expressed as the percentage increase in peak diameter.
Time Frame: Baseline and 4 weeks
Population: With the crossover design, participants completed both arms of the study with a two-week washout period in between.
Measure: Mean (Standard Deviation); unit: percentage of change in diameter
Arm/Group | Consumption of 100% Watermelon Juice | Consumption of a Placebo Beverage
Number analyzed (Participants) | 17 | 17
percentage of change in diameter | 2.85 (7.81) | 2.17 (9.25)

3. Primary Outcome: Change in Arterial Stiffness at 4 Weeks
Description: Determined by pulse wave velocity (PWV). A cuff-based system was used to measure brachial oscillometric pressure waveforms and generate central pressure curves by propriety algorithms. PWV was quantified as the rate at which a pulse wave moves down a vessel.
Time Frame: Baseline and 4 weeks
Population: With the crossover design, participants completed both arms of the study with a two-week washout period in between.
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Consumption of 100% Watermelon Juice | Consumption of a Placebo Beverage
Number analyzed (Participants) | 17 | 17
meters/second | -0.029 (0.269) | -0.188 (0.486)

ADVERSE EVENTS:
Time Frame: Four weeks for each intervention
Arm/Group | Consumption of 100% Watermelon Juice | Consumption of a Placebo Beverage
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-02-16): https://cdn.clinicaltrials.gov/large-docs/68/NCT03626168/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT03626168/ICF_001.pdf